CLINICAL TRIAL: NCT06063018
Title: A Single-arm, Single Center, Phase II Study of RC48 Combined With Tislelizumab for Second-line Treatment of HER2 Expression in Recurrent Cervical Cancer
Brief Title: RC48 Combined With Tislelizumab for Second-line Treatment of HER2 Expression in Recurrent Cervical Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K3956
Record Dates: First submitted 2023-09-11; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Cervical Cancer Recurrent
MeSH Terms: interventions — RC48 antibody; tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48 + Tislelizumab (Experimental): Durg：RC48: intravenous drip, 2mg/kg, D1, repeated once every 2 weeks. Durg ：Tislelizumab: intravenous drip, fixed dose 600 mg, D1, repeated once every 6 weeks.
  Interventions: Drug: RC48 + Tislelizumab

INTERVENTIONS:
Drug: RC48 + Tislelizumab — RC48: intravenous drip, 2mg/kg, D1, repeated once every 2 weeks. Tislelizumab: intravenous drip, fixed dose 600 mg, D1, repeated once every 6 weeks.

SUMMARY:
There is currently no standardized treatment for patients who have undergone first-line standard treatment. In this study, We investigated the efficacy and safty of RC48 combined with Tislelizumab in the second-line treatment of patients with HER2 expression in recurrent cervical cancer.

DETAILED DESCRIPTION:
This study is a single-arm, single center II study，aim to evaluate the effective and safe of RC48 combined with Tislelizumab in the second-line treatment of patients with HER2 expression in recurrent cervical cancer.

This study set up a safety introduction period, that is, the first 6 subjects enrolled in the study will be slowly monitored for safety. The monitoring time window was 28 days after first receiving the study drug. If Dose limit toxicity (DLT) is observed in ≥2 of the first 6 subjects and is assessed by the investigator team to be related to RC48 therapy, the initial dose of RC48 therapy in subsequent enrolled patients is adjusted to 1.5 mg/kg Q2W.

During the safety induction period, if a subject does not complete the safety assessment for the tolerability observation period (within 28 days after the first dose) for reasons other than dose tolerance, a new subject will be replaced.

After the safety introduction period, any enrolled subjects who withdraw early from the trial will not be allowed to be replaced by additional enrolled subjects. The number corresponding to the subject is not allowed to be reused by other new subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects aged from 18 to 75 years old；
2. Have Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0 or 1；
3. Have a life expectancy of at least 6 months, in the opinion of the investigator；
4. Histologically or cytologically confirmed primary cervical squamous cell carcinoma, adenocarcinoma, adenosquamous cell carcinoma, or small cell (neuroendocrine) cervical cancer;
5. Have measurable disease assessable by RECIST v1.1；
6. Adequate haematological, hepatic and renal functions defined by the protocol； Pathologically diagnosed patients with HER2 expression （defined as: IHC 3+ or IHC 2+ or HC 1+）advanced cervical cancer ；Note：It is also acceptable if the subject has previous test results (confirmed by the investigator)；
7. Negative blood pregnancy test at Screening for women of childbearing potential；Highly effective contraception for female subjects if the risk of conception exists；

Exclusion Criteria:

1. History of malignant tumors other than cervical cancer, except for the following two cases：a. The patient had received a potentially curative treatment and had no evidence of the disease for 5 years；b. Successful resection of skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder carcinoma, cervical carcinoma in situ, and other carcinoma in situ was received；
2. Previous malignant disease (other than cervical cancer) within the last 5 years with the exception of basal or squamous cell carcinoma of the skin or carcinoma in situ (bladder, cervical, colorectal, breast)Previous stem cell allogeneic or parenchymal organ transplants；
3. Patients who had previously received other anti-tumor systemic therapy (including traditional Chinese medicine with anti-tumor indications) less than 4 weeks before the use of this study, or adverse events caused by previous treatment did not recover to ≤CTCAE grade 1 (except for alopecia and pigmentation)；
4. Had received a live vaccine within 4 weeks prior to the start of study dosing or planned to receive any vaccine (except for COVID-19 vaccine) during the study period；
5. Previous or current congenital or acquired immunodeficiency disease；
6. Previous treatment with other antibody-coupled drugs；
7. Has not recovered from surgery, such as the presence of unhealed incisions or serious postoperative complications；
8. The patient had a known or suspected allergy to the experimental drug；
9. The New York College of Cardiology (NYHA) classiifies heart failure as grade 3 and above；
10. Severe infections that are active or poorly controlled clinically; Active infections, including: a. HIV (HIV1/2 antibody) positive; b. Active hepatitis B (HBsAg positive or HBV DNA > 2000IU/ml and abnormal liver function); c. Active hepatitis C (HCV antibody positive or ≥103 copies /ml of HCV RNA and abnormal liver function); d. active tuberculosis; d. Other uncontrolled active infections (CTCAE V5.0 > Grade 2);
11. Other significant clinical and laboratory abnormalities considered to affect safety assessment, such as uncontrolled diabetes, chronic kidney disease, grade II or above peripheral neuropathy (CTCAE V5.0), thyroid dysfunction, etc.； Other conditions deemed unsuitable for inclusion by the researchers；

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate（ORR） | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  Assess ORR, defined as Investigator-assessed CR + PR, per RECIST 1.1.

SECONDARY OUTCOMES:
Overall Survival(OS) | up to 3 years
  The time from the start of treatment with this study protocol to the time of all-cause death of patients.
Progression-free survival(PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  Time from initiation of study protocol treatment to disease progression (if occurring within 30 days of end of treatment) or death, as assessed by clinician or with or without radiographic progression.
Disease Control Rate (DCR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  Percentage of patients with CR/PR/SD in the number of patients that whose tumour can be evaluated.
Duration of response（DOR） | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  The time between the onset of efficacy and confirmation of tumor progression

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided